CLINICAL TRIAL: NCT07358195
Title: Addition of Venetoclax to Combined Reduced Intensity Hematopoietic Stem Cell and Kidney Transplantation for Patients With Chronic Kidney Disease and Hematologic Malignancy
Brief Title: Addition of Venetoclax to Combined Hematopoietic Stem Cell and Kidney Transplantation
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Thomas Spitzer, Professor of Medicine, Harvard Medical School Director Emeritus, Bone Marrow Transplant Program, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DFCC 25-668
Record Dates: First submitted 2026-01-05; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: Kidney Failure Chronic; Stem Cell Transplant; Stem Cell Transplant Complications; Tolerance; Hematologic Cancer
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hematologic Neoplasms | interventions — venetoclax; Kidney Transplantation; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Recipient (Experimental): Stem Cell and Kidney Transplant
  Interventions: Drug: Venetoclax; Procedure: Hematopoietic Cell Transplantation Conditioning Regimen; Procedure: Kidney Transplant; Procedure: Hematopoietic Cell Transplantation

INTERVENTIONS:
Drug: Venetoclax — Venetoclax 400mg orally once daily on days -8 through -1 with daily monitoring for tumor lysis syndrome. Venetoclax tablets will be swallowed (not crushed). Venetoclax dosing will not be repeated in the event of vomiting.
Procedure: Hematopoietic Cell Transplantation Conditioning Regimen — Cytoxan Day -6 & -5 Fludarabine Day -4, -3, -2 TBI Day -1
Procedure: Kidney Transplant — Living donor kidney transplant
Procedure: Hematopoietic Cell Transplantation — Donor bone marrow (target of 4 x 108 nucleated cells/kg of recipient ideal body weight)
  PBSC A goal dose of 5 x 106 CD34+ cells / kg of recipient actual body weight will be infused (minimum acceptable is 2 x 106 CD34+ cells / kg).

SUMMARY:
The primary objective is to assess the safety of the addition of venetoclax to reduced intensity conditioning for HLA-matched and haploidentical combined HSC and kidney transplantation as measured by stable full donor hematopoiesis and absence of CTCAE grade IV or V toxicity attributable to venetoclax.

ELIGIBILITY:
Recipient Inclusion Criteria:

* Patient ages 18-70
* Underlying hematological malignancy which is deemed as being potentially curable with allogeneic bone marrow or PBSC transplantation by the BMT voting team.
* Hematological malignancies include, but are not limited to: acute myeloid leukemia (AML), acute lymphoblastic leukemia (ALL), chronic myelogenous leukemia (CML), chronic lymphocytic leukemia (CLL), non-Hodgkin lymphoma (NHL), Hodgkin lymphoma, multiple myeloma (MM), myelodysplastic syndrome (MDS. Patient should be in a partial (PR) or complete remission (CR) at the time of the transplant.
* Existence of an HLA-matched or haploidentical relative who passes standard donor evaluations for bone marrow and kidney donation
* LVEF > 40% as measured by echocardiography or MUGA
* FEV1, FVC, and DLCO > 50% of predicted as measured by standard PFTs
* Total bilirubin < 2.0 (unless diagnosis of Gilbert's or hemolysis is made) and AST, ALT, alkaline phosphatase all < 5x institutions upper limit of normal
* ABO compatibility in the host vs. graft direction
* Men and women of reproductive potential must agree to use a reliable method of birth control during the treatment, and women should do so for a period of 1 year following the transplant.
* Participants should be on dialysis or have a CrCl ≤ 35 ml/min
* Life expectancy greater than 6 months
* Recipient ability to understand and provide informed consent

Donor Inclusion Criteria:

* HLA matched or haploidentical relative as defined by 3/6, 4/6, or 5/6 HLA-matched at HLA -A, -B, or -DRB1 who is 18-70 years of age
* ECOG performance status 0 or 1
* Excellent health per conventional pre-donor history (medical and psychosocial evaluation)

  • Acceptable laboratory parameters (hematology in normal or near-normal range; liver function < 3 times the upper limit of normal and normal creatinine)
* Compatible ABO blood group
* Negative donor lymphocyte cross match
* No positive testing for active viral infection (Hepatitis B, Hepatitis C, HIV)
* Donor ability to understand and provide informed consent
* Meets standard institutional criteria for both bone marrow or peripheral blood stem cell (PBSC) and kidney donation

Exclusion Criteria:

* Active serious infection
* Participation in other investigational drug use at the time of enrollment
* Positivity for active infection with HIV, HCV, or HBV
* ABO blood group incompatibility in the host-vs-graft direction

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of full donor chimerism | 24 months
Incidence of Grade IV Toxicity due to Venetoclax | Days -8 to Days -1
  NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Incidence of Grade V Toxicity due to Venetoclax | Days -8 to Days -1
  NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0

SECONDARY OUTCOMES:
Incidence of acute renal allograft rejection | 24 months
Incidence of delayed renal allograft rejection | 24 months
Incidence of acute GVHD | 24 months
Incidence of Chronic GVHD | 24 months
Patient Survival Rate | 24 months
Allograft Survival Rate | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States